CLINICAL TRIAL: NCT07157787
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of ALXN1920 in Adult Participants With PMN (Primary Membranous Nephropathy) Who Are at a High Risk for Disease Progression
Brief Title: Study of ALXN1920 in Adult Participants With Primary Membranous Nephropathy (PMN)
Acronym: AUTUMN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9900C00002; ALXN1920-PMN-201 (Other: Alexion); 2025-520780-40 (EudraCT Number)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Primary Membranous Nephropathy
Keywords: Primary Membranous Nephropathy; PMN; ALXN1920

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALXN1920 (Experimental): Participants will receive ALXN1920 subcutaneous (SC) and background treatment of ACE/ARB and Rituximab.
  Interventions: Drug: ALXN1920
- Placebo (Experimental): Participants will receive placebo subcutaneous (SC) and background treatment of ACE/ARB and Rituximab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALXN1920 — Participants will receive ALXN1920 SC infusion.
  Arms: ALXN1920
Drug: Placebo — Participants will receive Placebo SC infusion.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of ALXN1920 compared with placebo in participants with PMN who are at a high risk for disease progression using 24-hour urine protein creatinine ratio (UPCR).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a documented diagnosis of PMN, established by positive antiPLA2R antibody level (> 50 RU/mL) at Screening, which must be confirmed by a central laboratory
* Participants are willing to receive the background Standard of Care (SoC)
* Participants at high risk for disease progression, defined as:

  1. Receiving ACE inhibitor or ARB for a minimum of 8 weeks prior to Screening, with the dose titrated to the maximally tolerated level. Participants with less than 8 weeks on ACE inhibitor or ARB before Screening or who have not yet reached maximally tolerated dose will enter the Run-in Period.
  2. Participants who are on ACE inhibitor or ARB for a minimum of 8 weeks with Systolic Blood Pressure < 140 mmHg in ≥ 75% of the readings within last 8 weeks.
  3. Having two proteinuria measurements with each > 3.5 g/day, the second measurement showing ≤50% decrease from the first measurement.
* All participants must receive prophylactic treatment with appropriate antibiotics while receiving Rituximab (RTX), and be willing to be vaccinated against Neisseria meningitidis

Exclusion Criteria:

* Estimated glomerular filtration rate (GFR) < 60 mL/min/1.73 m^2 during Screening
* Documented rapid deterioration of kidney function
* History of life-threatening Nephrotic Syndrome within 1 year before Screening
* Diagnosis of anti- phospholipase A2 receptor (PLA2R) negative membranous nephropathy (MN) or anti-PLA2R positive MN but Screening serum anti-PLA2R < 50 RU/mL or kidney disease other than PMN
* History of kidney transplant or planned kidney transplant or dialysis during the Treatment Period
* History of other solid organ (heart, lung, small bowel, pancreas, or liver) or bone marrow transplant; or planned transplant during the Treatment Period
* History or presence of any clinically relevant co-morbidities
* History of intolerance or hypersensitivity to ACEi or ARB
* Use of SGLT2i, MRA, or ERA within 8 weeks prior to randomization and throughout the study period

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Proteinuria Based on 24-hour UPCR at Week 26 | Baseline, Week 26

SECONDARY OUTCOMES:
Change From Baseline in Proteinuria Based on 24-hour UPCR | Baseline
Change From Baseline in Proteinuria Based on Spot UPCR at Week 26 | Baseline and Week 26
Change From Baseline in Serum Albumin at Week 26 | Baseline and Week 26
Change From Baseline in Anti-phospholipase A2 Receptor (anti-PLA2R) Antibody Level at Week 26 | Baseline and 26
Change From Baseline in Peripheral Cluster of Differentiation 20 (CD20+) B Cell Count at Week 4, Week 8, and Week 26 | Baseline, Weeks 4, 8 and 26
Change From Baseline biomarker level at Week 26 | Baseline and Week 26

CONTACTS AND LOCATIONS:
Locations (37):
- United States (5):
  - Research Site, Loma Linda, California
  - Research Site, San Diego, California
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Houston, Texas
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
  - Research Site, Santa Fe
- Australia (3):
  - Research Site, Gosford
  - Research Site, Parkville
  - Research Site, Southport
- Brazil (3):
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
- China (4):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shenzhen
- France (3):
  - Research Site, Créteil
  - Research Site, Nice
  - Research Site, Toulouse
- Italy (3):
  - Research Site, Milan
  - Research Site, Ranica
  - Research Site, Torrette
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Toledo
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR